CLINICAL TRIAL: NCT00222040
Title: Microbubbles and Ultrasound in Stroke Trial: MUST Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: LLAU Marie-Elise, University Hospital Toulouse
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0302208
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2010-04-30 (Estimated); Status verified 2008-06

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke; thrombolysis; ultrasound; microbubbles; alteplase
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — High-Energy Shock Waves; SHU 508

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Levovist
  Interventions: Radiation: Ultrasound; Drug: Levovist
- 2 (No Intervention): No specific intervention

INTERVENTIONS:
Radiation: Ultrasound — 2-MHz, low intensity transcranial ultrasound
  Arms: 1
Drug: Levovist — D-Galactose and palmitic palmitique intravenous 4 g
  Arms: 1

SUMMARY:
To determine whether transcranial 2-MHz ultrasound combined with intravenous administration of microbubbles improves early recanalization in patients with acute ischemic stroke caused by middle cerebral artery (MCA) proximal occlusion treated with intravenous alteplase within 3 hours of symptom onset.

DETAILED DESCRIPTION:
Proximal MCA occlusion is recognized using MR or CT angiography performed before inclusion. All patients are treated with alteplase according to current guidelines. In addition, patients randomized in the active group are continuously exposed to transcranial 2-MHz ultrasound for 1 hour combined with intravenous administration of microbubbles. Controls are only treated with alteplase. The ultrasound beam is positioned at the thrombus/blood flow interface using color-coded sonography. Galactose-based microbubbles are administered via continuous intravenous infusion over 40 min.

Early recanalization is assessed using MR or CT angiography 4 to 8 hours after symptom onset. The evaluation of angiograms is performed by 2 neuroradiologists blinded to group of randomization and clinical details. The primary outcome measure is the rate of early recanalization. Recanalization is assessed using the TIMI classification. Secondary endpoints include the rate of symptomatic intracerebral hemorrhage, mortality, and functional outcome on the modified Rankin scale at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke
* MCA proximal occlusion on CT or MR angiography
* Thrombolysis with intravenous alteplase initiated within 3 hours of stroke onset

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-06; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Rate of early recanalization on post-treatment MR or CT angiography. Recanalization is described using the tIMI classification.

SECONDARY OUTCOMES:
Rate of symptomatic intracerebral hemorrhage, mortality, Score on the modified Rankin scale | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: LARRUE Vincent, MD, Principal Investigator — University Hospital, Toulouse, France
Locations (5):
- France (5):
  - Service de Neurologie, Besançon
  - Service de Neurologie, Hôpital Gui de Chauliac, Montpellier
  - Service de Neurologie, Hôpital Sainte Anne, Paris
  - Service de Neurologie Vasculaire, University Hospital, Toulouse
  - Service de Neurologie, University Hospital, Tours

REFERENCES:
- [Background] Cintas P, Le Traon AP, Larrue V. High rate of recanalization of middle cerebral artery occlusion during 2-MHz transcranial color-coded Doppler continuous monitoring without thrombolytic drug. Stroke. 2002 Feb;33(2):626-8. doi: 10.1161/hs0202.103073. PMID 11823681
- [Background] Cintas P, Nguyen F, Boneu B, Larrue V. Enhancement of enzymatic fibrinolysis with 2-MHz ultrasound and microbubbles. J Thromb Haemost. 2004 Jul;2(7):1163-6. doi: 10.1111/j.1538-7836.2004.00746.x. PMID 15219200
- [Background] Viguier A, Petit R, Rigal M, Cintas P, Larrue V. Continuous monitoring of middle cerebral artery recanalization with transcranial color-coded sonography and Levovist. J Thromb Thrombolysis. 2005 Feb;19(1):55-9. doi: 10.1007/s11239-005-0940-6. PMID 15976968